CLINICAL TRIAL: NCT04332406
Title: Normal Ventilatory and Perfusion Pulmonary Function in TEMP: Generation of 3D Statistical Maps From Normal Examinations
Brief Title: Normal Ventilatory and Perfusion Pulmonary Function in TEMP
Acronym: 3DSPECSTAT
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0129
Record Dates: First submitted 2019-09-26; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Patents With Normal VQ/SPECT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ventilation - perfusion SPECT is attractive for lung function assessement. Unfortunately, it is very difficult to delineate normal to abnormal areas because of physiological uptake heterogeneity.

In that context, it would be of interest to build statistical maps from registrered normal studies and propose a new methodology for normal SPECT delineation

DETAILED DESCRIPTION:
Patients with normal VQ SPECT-CT will be analysed. After a image proccesing workflow including rigid registration, non rigid registration and normalization, a voxelized mean and standard deviation map will be created. Those maps will be analyzed in regards of physiology and litterature.

ELIGIBILITY:
Inclusion Criteria:

* normal perfusion and ventilation scans, and no parenchyma or pleural abnormality on low dose CT
* confirmation by a second senior physician

Exclusion Criteria:

Patients with history of pulmonary disease:

* chronic obstruction pulmonary disease,
* previous pulmonary embolism,
* surgery of the lungs
* radiotherapy of the lungs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the department of nuclear medicine of Brest University Hospital, France, for suspected acute pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Posterior to Anterior and Inferior to Superior uptake relative difference on parametric mean registered SPECT map versus non registered SPECT | through study completion, an average of 3 months
  parametric mean and standard deviation maps are build from elastic registration of normal lung V/Q SPECT-CT. A ROI based quantitative regional uptake comparison is performed to verify the influence of elastic registration on radiotracer distribution

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Yves Le Roux, MD, Phd, Study Director — CHRU Brest
Locations (1):
- Médecine nucléaire - Hôpital Morvan (CHRU de Brest), Brest, France